CLINICAL TRIAL: NCT07160179
Title: Safety, Tolerability, Pharmacokinetics, and Exploratory Efficacy of ABBV-6628 in Subjects With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Brief Title: Study to Assess the Adverse Events and How Intravitreal ABBV-6628 Moves Through the Body of Adult Participants With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M24-204
Record Dates: First submitted 2025-08-12; First posted 2025-09-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Geographic Atrophy; Age-Related Macular Degeneration
Keywords: Geographic Atrophy; Age-Related Macular Degeneration; ABBV-6628
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- ABBV-6628: Stage 1-Cohort 1 (Experimental): Participants will receive a single dose of ABBV-6628 in Cohort 1 on day 1.
  Interventions: Drug: ABBV-6628
- ABBV-6628: Stage 1 -Cohort 2 (Experimental): Participants will receive a single dose of ABBV-6628 in Cohort 2 on day 1.
  Interventions: Drug: ABBV-6628
- ABBV-6628: Stage 1 -Cohort 3 (Experimental): Participants will receive a single dose of ABBV-6628 in Cohort 3 on day 1.
  Interventions: Drug: ABBV-6628
- ABBV-6628: Stage 1 -Cohort 4 (Experimental): Participants will receive ABBV-6628 in Cohort 4 on day 1 and month 2.
  Interventions: Drug: ABBV-6628
- ABBV-6628: Stage 2 (Experimental): Participants will receive ABBV-6628 for approximately 22 months followed by 3 months of follow-up.
  Interventions: Drug: ABBV-6628
- SYFOVRE: Stage 2 (Experimental): Participants will receive SYFOVRE for approximately 22 months followed by 3 months of follow-up.
  Interventions: Drug: SYFOVRE

INTERVENTIONS:
Drug: ABBV-6628 — Intravitreal injection
  Arms: ABBV-6628: Stage 1 -Cohort 2; ABBV-6628: Stage 1 -Cohort 3; ABBV-6628: Stage 1 -Cohort 4; ABBV-6628: Stage 1-Cohort 1; ABBV-6628: Stage 2
Drug: SYFOVRE — Intravitreal injection
  Arms: SYFOVRE: Stage 2

SUMMARY:
Age-related macular degeneration (AMD) is the abnormal growth of new blood vessels in the light-sensitive tissue at the back of the eye called the retina. Geographic Atrophy (GA) is an advanced form of dry AMD. The purpose of this study is to assess the adverse events and how intravitreal ABBV-6628 moves through the body of adult participants with secondary to age-related macular degeneration

ABBV-6628 is an investigational monoclonal antibody fragment being developed for the treatment of geographic atrophy (GA) secondary to (AMD) age-related macular degeneration. Participants in the Stage 1 part will be placed in 1 of 4 groups, called treatment arms. Participants in Stage 2 will be placed into 1 of 2 groups. Each group receives different treatment. Adult participants aged 50 and older years with a diagnosis GA secondary to age-related macular degeneration will be enrolled. Around 66 participants will be enrolled in the study at approximately 27 sites across the US.

Participants in Stage 1 will be given ABBV-6628 as an intravitreal injection (injection into the jelly-like tissue that fills the eyeball injection) with dose escalation. Participants in Stage 2 will receive ABBV-6628 or SYFOVRE, an approved treatment for geographic atrophy, administered as per the FDA-approved label. The treatment duration is approximately 22 months and 3 months of follow-up.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular weekly visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Stage 1 and Stage 2

-Diagnosed with Geographic atrophy (GA) secondary to age-related macular degeneration (AMD) in the study eye.

Stage 1

* Foveal or non-foveal GA with total GA lesion area ≥ 0.5 DA (1.25 mm2) in the study eye, as assessed by the investigator at Screening and confirmed by the central reading center prior to Baseline/Day 1
* Absence of choroidal neovascularization (CNV) in the study eye as assessed by the investigator at Screening and confirmed by the central reading center prior to Baseline/Day 1. In addition, investigators should confirm eligibility prior to treatment administration on Baseline/Day 1.

Stage 2

* Non-foveal GA with total lesion area of 1 to 7 DA (2.5 to 17.5 mm2); within 0.5 to 1.5 mm from fovea center in the study eye, as assessed by the investigator at Screening and confirmed by the central reading center prior to Baseline/Day 1.
* Absence of CNV in both eyes as assessed by the investigator at Screening and confirmed by the central reading center prior to Baseline/Day 1. In addition, investigators should confirm eligibility prior to treatment administration on Baseline/Day 1.

Exclusion Criteria:

Stage 1 and Stage 2

* History of recurrent or currently active ocular or intraocular inflammation (e.g., uveitis, endophthalmitis) in at least one eye at Screening and Baseline/Day 1.
* Active periocular, ocular, or intraocular infection in at least one eye at Baseline/Day 1.
* History or clinical signs of diabetic retinopathy, diabetic macular edema (DME), or any retinal vascular disease other than AMD in at least one eye at Screening and Baseline/Day 1.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to approximately 25 months
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Number of Participants with Abnormal Change in Physical Examinations | Up to approximately 25 months
  Number of participants with abnormal change in physical examinations in areas like cardiovascular, respiratory, gastrointestinal, and neurological systems will be assessed.
Number of Participants with Abnormal Change From Baseline in Vital Sign Measurements | Up to approximately 25 months
  Number of participants with abnormal change from baseline in vital sign measurements like systolic and diastolic blood pressure will be assessed.
Change From Baseline in Electrocardiograms (ECGs) | Up to approximately 25 months
  12-lead resting ECGs will be recorded. Parameters include heart rate, PR interval, QT interval, QRS duration, and QT interval corrected using Fridericia's formula (QTcF).
Number of Participants with Abnormal Change in Clinical Laboratory Test Results Like Hematology will be Assessed | Up to approximately 25 months
  Number of participants with abnormal change in clinical laboratory test results like hematology will be assessed.
Change from baseline in Best Corrected Visual Acuity (BCVA) | Up to approximately 25 months
  BCVA measured by Early Treatment Diabetic Retinopathy Study (ETDRS) (normal luminance and low luminance visual acuity)
Change in Slit lamp biomicroscopy assessment | Up to approximately 25 months
  Changes in Slit lamp biomicroscopy assessed by the physician will be assessed.
Change in Intraocular pressure (IOP) | Up to approximately 25 months
  Measured by using Goldmann applanation tonometry (GAT) or hand-held tonometer
Change in Lens examination assessment | Up to approximately 25 months
  Changes in Lens examination assessed by the physician will be assessed.
Change in Ophthalmoscopy assessment | Up to approximately 25 months
  Changes in Ophthalmoscopy assessed by the physician will be assessed.
Change in fundus autofluorescence (FAF) imaging assessed by Investigator | Up to approximately 25 months
  Fundus autofluorescence (FAF) imaging assessed by Investigator
Change in Retinal evaluation | Up to approximately 25 months
  Measured by color fundus photography (CFP) imaging assessed by Investigator
Change in spectral domain optical coherence tomography (SD-OCT) | Up to approximately 25 months
  Spectral domain optical coherence tomography (SD-OCT)
Change in Fluorescein angiography (FA) assessed by Investigator. | Up to approximately 25 months
  Fluorescein angiography (FA) assessed by Investigator
Change in choroidal neovascularization (CNV) assessed by Investigator. | Up to approximately 25 months
  Choroidal Neovascularization (CNV) assessed by Investigator.
Percentage of Participants with Clinically Significant Post-treatment Administration Assessment (study eye only) Findings as Assessed by the Investigator | Up to approximately 25 months
  Post-treatment Administration Assessment (study eye only)
Maximum Serum Concentration (Cmax) of ABBV-6628 | Up to approximately 25 months
  Cmax of ABBV-6628
Time to Cmax (Tmax) of ABBV-6628 | Up to approximately 25 months
  Tmax of ABBV-6628
Area Under the Concentration-Time Curve From zero to the last measurable Timepoint (AUC0-Tlast) of ABBV-6628 | Up to approximately 25 months
  AUC0-Tlast of ABBV-6628
Stage 2-Trough serum concentration immediately before next dose (Ctrough) of ABBV-6628 | Up to approximately 12 months
  Ctrough of ABBV-6628

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- United States (4):
  - Retina Partners Midwest, P.C. /ID# 262172, Carmel, Indiana
  - Retina Research Institute of Texas /ID# 262141, Abilene, Texas
  - Retina Foundation of the Southwest /ID# 262479, Dallas, Texas
  - Retina Consultants - The Woodlands /ID# 262138, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-204